CLINICAL TRIAL: NCT06798753
Title: The Presence of Ureteral Calculi Upon Supine PCNL Completion: Occlusion Balloon Catheter Versus 5FR Ureteral Catheter
Brief Title: Occlusion Balloon vs. 5FR Ureteral Catheter
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Mantu Gupta, Chair of Urology, MSW and MSM Hospitals Professor, Icahn School of Medicine at Mount Sinai Director of Endourology, Mount Sinai Medical Center Editor-in-Chief, Videourology, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: STUDY-24-01650
Record Dates: First submitted 2025-01-23; First posted 2025-01-29 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Kidney Stones
Keywords: percutaneous nephrolithotomy; PCNL; Occlusion Balloon Catheter; kidney stone
MeSH Terms: conditions — Kidney Calculi

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Occlusion Balloon Catheter (Active Comparator): The occlusion balloon catheter (OBC) is a type of ureteral catheter equipped with a small inflatable balloon at its tip. When inflated, the balloon can help prevent the migration of stone fragments.
  Interventions: Device: Occlusion Balloon Catheter
- 5FR Ureteral Catheter (Active Comparator): The 5FR ureteral catheter (5FR-UC) is an open-ended small-caliber tube inserted at the beginning of PCNL to facilitate visualization of the collecting system using fluoroscopy and assist with renal access.
  Interventions: Device: 5FR Ureteral Catheter

INTERVENTIONS:
Device: Occlusion Balloon Catheter — The occlusion balloon catheter (OBC) is a type of ureteral catheter equipped with a small inflatable balloon at its tip. When inflated, the balloon can help prevent the migration of stone fragments.
  Arms: Occlusion Balloon Catheter
Device: 5FR Ureteral Catheter — The 5FR ureteral catheter (5FR-UC) is an open-ended small-caliber tube inserted at the beginning of PCNL to facilitate visualization of the collecting system using fluoroscopy and assist with renal access.
  Arms: 5FR Ureteral Catheter

SUMMARY:
Occlusion Balloon catheter provides the ability to occlude the exit of the kidney pelvis during percutaneous nephrolithotomy (PCNL) and potentially prevents the migration of stone fragments into the ureter. The necessity for it might be questioned during supine PCNL due to the upward oblique position of the kidney. The objective of the study is to compare the presence of ureteral stone fragments upon completion of supine PCNL with and without using an occlusion balloon catheter (OBC).

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years and older.
* Diagnosed with kidney stones and scheduled for PCNL.
* Able and willing to provide informed consent.

Exclusion Criteria:

* Pregnant women
* Urinary tract anomalies such as urinary diversion, previous ureteral reconstruction surgeries, horseshoe kidney, solitary kidney, duplicated system, urinary stricture disease, ureteropelvic junction obstruction, pelvic kidney, stone in calyceal diverticulum.
* Prone procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2025-01-23 (Actual); Primary Completion 2025-08-29 (Actual); Study Completion 2025-08-29 (Actual)

PRIMARY OUTCOMES:
Number of ureteral stone fragments identified endoscopically | During procedure
  Endoscopic identification of ureteral stone fragments will be used to compare rate of ureteral stone fragments upon completion of PCNL while using OBC versus 5FR-UC.

SECONDARY OUTCOMES:
Length of procedure | During procedure
  Length of procedure is a common procedural outcome of endourologic procedures.

CONTACTS AND LOCATIONS:
Overall Officials: Mantu Gupta, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai West, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Results will be shared in aggregate to protect subject privacy

DOCUMENTS (1):
  • Informed Consent Form (2025-12-15): https://cdn.clinicaltrials.gov/large-docs/53/NCT06798753/ICF_000.pdf